CLINICAL TRIAL: NCT00297986
Title: Evaluation of Different Interfaces for NPPV
Brief Title: Evaluation of Different Interfaces for Noninvasive Positive Pressure Ventilation (NPPV)
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 1040
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Respiratory Failure; Healthy
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Head Protective Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: healthy subjects
  Interventions: Device: Helmet

INTERVENTIONS:
Device: Helmet — Evaluation of different interfaces for NPPV

SUMMARY:
In this study the investigators aimed to study the ventilatory performance of different interfaces during NPPV delivering.

DETAILED DESCRIPTION:
We will test the ventilatory performance in term of ventilatory pattern, muscle effort and gas exchange of different interfaces for NPPV.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy subjects

Exclusion Criteria:

* Barotrauma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy